CLINICAL TRIAL: NCT03598062
Title: Knowledge , Attitudes and Educational Experiences of A Group of Egyptian Dental Students Regarding Physical Child Abuse :A Cross Sectional Study
Brief Title: Knowledge,Attitudes and Eductional Experiences of a Group of Egyptian Dental Students Regarding Physical Chid Abuse
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Ibrahim Ahmed, Dentist, Cairo University
Other Study IDs: CEBD-CU-2018-06-28
Record Dates: First submitted 2018-07-01; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Conditions Child Abuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

SUMMARY:
Scientific background ( Statement of the problem) :

Child abuse continues to be a serious social problem amongst all cultural and socio-economic groups that causing physical and emotional trauma to children and can even lead to death. Child abuse or child maltreatment is physical, sexual or psychological maltreatment or neglect of a child, especially by a parent or caregiver. The term child abuse and child maltreatment are used interchangeably ( WHO,2002 ) . Although the Egyptian child law no.12 of 1996 saves the right of the child to life, survival, and development in a supportive family environment and to be protected from all forms of violence, or injury, or physical, mental or sexual abuse Egyptian children facing different types of abuse (UNICEF Egypt,2014) .

Dentists are in the most favourable position to recognise child abuse , because 50-75 % of reported lesions involve the mouth region, the face and the neck but many dentists fail to report suspected cases of abuse ( Bodrumlu et al.,2016 and Kaur et al.,2017 ) . The quality of dental education could be one crucial factor that may contribute to an increase in the detection and the reporting of child maltreatment by dental care providers and students (Malpani et al. ,2017) .

Rationale for carrying out this study As there is no sufficient data about Egyptian dental students's knowledge and attitude in regard to child physical abuse , so the aim of this study is to assess the knowledge, attitudes and educational experiences of a group of Egyptian dental students regarding child physical abuse .

Benefits to the practitioners

* Increase the awareness of dental students about child abuse and their role in child protection.
* Discovering the main reasons for not reporting suspicion of child abuse.
* Knowledge about physical signs of abuse will help dental students in detecting child abuse cases.

Benefits to the patient and population

* Increase the knowledge and awareness of all health care providers toward child abuse will help in detection of child abuse cases and child protection .
* Asking the parents or care giver about the physical signs that may indicate child abuse will make them fear from reporting and stop their act.

DETAILED DESCRIPTION:
Review of literature Databases and websites as PubMed, Google scholar were searched for relevant literature until October 2017 with key words "Child abuse, Child maltreatment, Physical child abuse, Violence against children, Dental students " .

Thomas et al., 2006 conducted a study to explore dental and dental hygiene students' educational experiences and knowledge toward child abuse. Data were collected by 233 dental (116 male/117 female) and 76 female dental hygiene students at the University of Michigan through a self -administrated questionnaire. The results showed that 94.7 %of the dental hygiene and 70.5 % of the dental students reported having learned about child abuse in classroom settings, and 15.8 %of the dental hygiene and 29.3 % of the dental students reported having learned about it in clinical settings .Only 5.5% of the dental and 16.7 %of the dental hygiene students defined child abuse correctly; 32.2 %of the dental and 13.2 %of the dental hygiene students did not know their legal responsibility concerning reporting child abuse and 82.4% of the dental and 78.9% of the dental hygiene students did not know where to report child abuse. Dental and dental hygiene curricula should be improved to ensure that students are well prepared for their role in child protection.

Al-Jundi et al., 2010 conducted a study to assess eductional experiences ,attitude and knowledge of Jordanian dental students toward child physical abuse. Data were collected through a self-administered questionnaire completed by 441 undergraduate and postgraduate dental students in both dental schools in Jordan. study indicated that both undergraduate and postgraduate dental students are not sufficiently prepared to undergo their role in protection of children from abuse.

Jordan et al., 2012 conducted a study to assess the educational experiences and knowledge of a group of Croatian dental students regarding child abuse and neglect. Questionnaires were completed by 544 students (153 male &391 female) from all six years at the University of Zagreb School of Dental Medicine with a response rate of 74.9%. The results indicate lack of knowledge of the signs of physical and sexual abuse of children. Students from more senior teaching years have a greater amount of knowledge related to child abuse and neglect compared to students from more junior teaching years. In conclusion, dental students should be better educated and prepared for their important role in protecting children from abuse .

Hashim et al., 2013 conducted a study to assess educational experience, attitudes and knowledge toward child physical abuse among a group of dental students in United Arab Emirates. a self-administered structured questionnaire completed by 578 under graduate dental students ,The results indicated that there was lack of knowledge of reporting procedure, signs of physical abuse and social indicators among all participants. Over 80 % of the students agreed that dentists should report abuse cases and 94.3 % of the participants believed they had an ethical duty to report child abuse. Most students indicated that their dental school was the main source of information on child physical abuse. The majority of the respondents expressed a need for further training.

Hazar Bodrumlu et al., 2016 conducted a study to assess dental students' knowledge and attitudes towards child abuse at the Faculty of Dentistry of the Ondokuz Mayis University. The data were collected through a self-report questionnaire administered completed by dental students (137 female/111 male) in three different dental classes (third, fourth and fifth study years) with 100 % response rate. About 67.74% of the third year, 40.71% of the fourth year and 16.67% of the fifth year believed that they could detect child abuse cases. However, there is a lack of knowledge of social indicators, signs of physical abuse and reporting procedure amongst all participants. The assessment of the total correct answers indicate significant differences amongst third-, fourth- and fifth-year students' answers. Fifth-year students had the highest rate of correct responses (P < 0.05). Most students wanted to receive more knowledge about child abuse.

Aim of the study :

The aim of this study is to:

assess knowledge ,attitude and educational experiences of a group of Egyptian dental students regarding physical child abuse.

PO:

(P) Population: dental students (3rd to 5th classes) from Faculty of Dentistry ,Cairo University.

(O) Outcomes :Knowledge, attitude, educational experience of dental students toward physical child abuse.

Research question What is the knowledge ,attitude and educational experiences about physical child abuse among a group of Egyptian dental students(3rd to 5th classes) from Faculty of Dentistry ,Cairo University ? Study design: Cross-sectional study.

Study settings:

* Questionnaires ,Appendix 1will be distributed to the students and give them 30 minutes to answer it.
* All questionnaires will be collected at the same day, to prevent any of the participants to search for the answers of questions that related to their knowledge.
* Participants during answering the questionnaire are not allowed to ask their colleagues, to ensure accuracy of the answers of knowledge questions.
* The researcher is not allowed to help the participant in answering the questions.
* Participants are allowed to ask the researcher any question either to clarify any part of the questions or anything about the survey.
* The researcher will deal with the participant personally, so there is no risk of the same dentist to complete more than one questionnaire.

After the participants finish answering the questionnaires, it will be collected and subjected to data analysis.

Study size:

the investigator is going to apply a convenient consecutive sampling ;it will include all dental students (3rd to 5th classes) at faculty of Dentistry ,Cairo University. Students will be invited to complete the questionnaire. All number of students will be reported , response rate will be calculated and no attempt is made to follow up with dentists who were absent in the day of the survey.

Statistical methods:

The data will be analyzed using the statistical analysis software SPSS version 20.the individual scores will be summed up to the yield total score. Descriptive statistic will be calculated as mean scores,standar deviation and frequency distribution.

The difference of knowledge ,personal views and experiences betwwen different categories will be assessed by students t-test or ANOVA according to the number of categories .

The difference between male and females doctors will be assessed by students t-test. P value <0.05 will be considered significant : All test will be two tails.

Ethical consideration

* A permission letter, explaining the aim of the study will be presented to the Pediatric Dentistry and Dental Public Health Department Head - Cairo University granting approval to conduct this survey among faculty of dentistry students.
* An informed consent explaining the aim of the study will be signed by the participants.

ELIGIBILITY:
Inclusion Criteria:

- 1.Egyptian dental students (3rd to 5th ) classes in Faculty of Dentistry ,Cairo University.

2.Both genders are included

Exclusion Criteria:

* Dental students who refuse to participate in the study .

Ages: 19 Years to 25 Years | Sex: All
Age Groups: Adult
Gender Based: Yes
Study Population: All Egyptian dental students (3rd to 5th ) classes in Faculty of Dentistry ,Cairo University
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Knowledge, attitude, educational experience of dental students toward physical child abuse | 3 monthes
  Measuring unit Structured self-administered questionnaire (Al-Jundi et al .,2010, Jordan et al.,2012 , Hashim et al., 2013 and Hazar Bodrumlu et al.,2016) measuring units :Numbers and percentages (The questionnaire include binary and MCQ)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Jundi SH, Zawaideh FI, Al-Rawi MH. Jordanian dental students' knowledge and attitudes in regard to child physical abuse. J Dent Educ. 2010 Oct;74(10):1159-65. PMID 20930248
- [Background] Hashim R, Al-Ani A. Child physical abuse: assessment of dental students' attitudes and knowledge in United Arab Emirates. Eur Arch Paediatr Dent. 2013 Oct;14(5):301-5. doi: 10.1007/s40368-013-0063-2. Epub 2013 Jul 4. PMID 23824733
- [Background] Hazar Bodrumlu E, Avsar A, Arslan S. Assessment of knowledge and attitudes of dental students in regard to child abuse in Turkey. Eur J Dent Educ. 2018 Feb;22(1):40-46. doi: 10.1111/eje.12242. Epub 2016 Oct 13. PMID 27735105
- [Background] Jordan A, Welbury RR, Tiljak MK, Cukovic-Bagic I. Croatian dental students' educational experiences and knowledge in regard to child abuse and neglect. J Dent Educ. 2012 Nov;76(11):1512-9. PMID 23144487
- [Background] Kaur H, Vinod KS, Singh H, Arya L, Verma P, Singh B. Child maltreatment: Cross-sectional survey of general dentists. J Forensic Dent Sci. 2017 Jan-Apr;9(1):24-30. doi: 10.4103/jfo.jfds_6_15. PMID 28584471
- [Background] Malpani S, Arora J, Diwaker G, Kaleka PK, Parey A, Bontala P. Child Abuse and Neglect: Do We know enough? A Cross-sectional Study of Knowledge, Attitude, and Behavior of Dentists regarding Child Abuse and Neglect in Pune, India. J Contemp Dent Pract. 2017 Feb 1;18(2):162-169. doi: 10.5005/jp-journals-10024-2009. PMID 28174372
- [Background] Thomas JE, Straffon L, Inglehart MR. Child abuse and neglect: dental and dental hygiene students' educational experiences and knowledge. J Dent Educ. 2006 May;70(5):558-65. PMID 16687641